CLINICAL TRIAL: NCT05083013
Title: Outcomes of Diabetes In Hospitalized COVID-19 Patients At Assiut University Hospital
Brief Title: Diabetes In Relation to Hospitalized COVID-19 Patents At Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Martina Saad Lamey, Principal Investigator, Assiut University
Other Study IDs: outcomes of DM in COVID-19
Record Dates: First submitted 2021-10-10; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus; COVID-19
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 with DM: All patients will be screened for diabetes according to history and blood glucose measurements as well as HbA1C.
  Accordingly, the patients will be divided into two groups, diabetic and non-diabetic group.
  Interventions: Diagnostic Test: Reverse transcription polymerase chain reaction (RT-PCR); Diagnostic Test: Glycated haemoglobin (HbA1C); Radiation: High Resolution Computed Tomography (HRCT); Diagnostic Test: Routine Laboratory investigations; Diagnostic Test: Random Blood Sugar (RBS)
- COVID-19 without DM: All patients will be screened for diabetes according to history and blood glucose measurements as well as HbA1C.
  Accordingly, the patients will be divided into two groups, diabetic and non-diabetic group.
  Interventions: Diagnostic Test: Reverse transcription polymerase chain reaction (RT-PCR); Diagnostic Test: Glycated haemoglobin (HbA1C); Radiation: High Resolution Computed Tomography (HRCT); Diagnostic Test: Routine Laboratory investigations; Diagnostic Test: Random Blood Sugar (RBS)

INTERVENTIONS:
Diagnostic Test: Reverse transcription polymerase chain reaction (RT-PCR) — For SARS Corona Virus 2 (COV2) confirmation
  Other Names: Reverse transcription polymerase chain reaction
Diagnostic Test: Glycated haemoglobin (HbA1C) — Diabetic patients' group will be categorized according to their glycemic control by using their glycated haemoglobin (HBA1C) into good control, fair control and poor control
  Other Names: Glycated haemoglobin
Radiation: High Resolution Computed Tomography (HRCT) — with the coronavirus disease 2019 Reporting and Data System (CO-RADS) classification grade 5 for SARS COV2 confirmation
  Other Names: High Resolution Computed Tomography
Diagnostic Test: Routine Laboratory investigations — * Arterial blood gases (ABGs)
  * Routine Laboratory investigations (Urea, Creatinine, Liver function tests, Serum Electrolytes, Prothrombin Concentration)
Diagnostic Test: Random Blood Sugar (RBS) — Blood Sugar will be measured before each meal and before bed time during hospitalization.

SUMMARY:
Coronavirus disease (COVID-19), a global pandemic affecting the whole world and taking the lives of millions. The majority of fatalities occur in the elderly specially in the presence of chronic diseases such as diabetes mellitus (DM), hypertension, obesity, cardiovascular disease, chronic kidney disease and cancer.

DETAILED DESCRIPTION:
Knowing about the family of coronaviruses is that they are the cause of a variety of well-known diseases affecting humans, ranging from common cold to the Middle East Respiratory Syndrome (MERS) and Acute Severe Respiratory Syndrome (SARS), and now the COVID-19 as a new problematic family member.

Regarding DM as a knowing old health problem, it has been found that we can use it in predicting the prognosis of the COVID-19 as admission to intensive care unit, invasive ventilation or even death.

Previous studies confirmed that uncontrolled DM can badly affects innate immunity which considered as the first line of defence mechanism against COVID-19 infection.

In addition, DM has a pro-inflammatory effect through exaggeration of cytokine response which appears clearly through higher results of serum levels of interleukin-6 (IL-6), C-reactive protein and ferritin, this suggests that people with DM are more venerable to cytokine storm which leads to Acute Respiratory Distress Syndrome (ARDS), shock and rapid deterioration of the case.

On the other hand, on looking to previous studies and data collected about the prior SARS outbreak in 2003, which suggested that COVID-19 can lead to worsening of glycemic control in known diabetic patients and above that caused by the stressful nature of a critical illness.

In addition, COVID-19 can lead to increasing insulin resistance specially in patients with type II DM. Also, the medications used in the management of COVID-19 having an indirect role on worsening of blood sugar levels also should be taken in our consideration, Corticosteroids as an example, used in the management of patients having ARDS or sepsis can lead to changes in their glycemic profile.

ELIGIBILITY:
Inclusion Criteria:

* Cases aged 18 years and over.
* Cases diagnosed as COVID-19 positive.
* Cases admitted to Assiut University Hospitals.

Exclusion Criteria:

* Age less than 18 years.
* Outpatient management (even in confirmed cases of COVID-19).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to Assiut University Hospital from the 1st of Oct. 2021 to 1st of Oct. 2022 with confirmed COVID-19 infection, will be included, based on WHO case definitions of COVID-19 All patients will be surveyed and scored by the criteria of COVID-19 severity index, and accordingly categorized into low, moderate, high and critically ill cases All patients will be screened for DM according to history and blood glucose measurements as well as HbA1C.
  Accordingly, the patients will be divided into two groups, diabetic and non-diabetic group.
  Diabetic patients' group will be categorized according to their glycemic control by using their glycated hemoglobin (HBA1C) used to determine their past two to three-month glycemic control, into good control, fair control and poor control
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rates | up to 1 year
  mortality rate among diabetic and non diabetic COVID-19 patients
Hospital stays | up to 1 year
  for how long patients admitted to hospital
Need for ICU admission | up to 1 year
  who will need ICU admission during patient hospitalization
Need for ventilatory support | up to 1 year
  who will need for ventilatory support (Non-Invasive ventilation (NIV), High Flow Nasal Cannula (HFNC) and Invasive Mechanical Ventilation (IMV).

SECONDARY OUTCOMES:
Glycemic control | up to 1 year
  monitoring of glycemic control among patient groups
Newly onset DM will appear among non-diabetic patients | up to 1 year
  who will develop DM among non-diabetic group
Acute complications of diabetes | up to 1 year
  as hypoglycaemia, diabetic ketoacidosis and hyperosmolar nonketotic coma
Exacerbation of chronic complications of diabetes | up to 1 year
  as diabetic retinopathy, nephropathy and neuropathy
Changes of diabetes management plan | up to 1 year
  who will be shifted from oral to insulin therapy and who will be changed of their insulin regimen or introduction form from subcutaneous to intravenous infusion
Incidence of other complications | up to 1 year
  as hypertension renal and liver diseases

CONTACTS AND LOCATIONS:
Overall Officials: Martina S. Lamey Eskander, MBBCH., Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Result] Guan WJ, Liang WH, Zhao Y, Liang HR, Chen ZS, Li YM, Liu XQ, Chen RC, Tang CL, Wang T, Ou CQ, Li L, Chen PY, Sang L, Wang W, Li JF, Li CC, Ou LM, Cheng B, Xiong S, Ni ZY, Xiang J, Hu Y, Liu L, Shan H, Lei CL, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Cheng LL, Ye F, Li SY, Zheng JP, Zhang NF, Zhong NS, He JX; China Medical Treatment Expert Group for COVID-19. Comorbidity and its impact on 1590 patients with COVID-19 in China: a nationwide analysis. Eur Respir J. 2020 May 14;55(5):2000547. doi: 10.1183/13993003.00547-2020. Print 2020 May. PMID 32217650
- [Result] Jafar N, Edriss H, Nugent K. The Effect of Short-Term Hyperglycemia on the Innate Immune System. Am J Med Sci. 2016 Feb;351(2):201-11. doi: 10.1016/j.amjms.2015.11.011. PMID 26897277
- [Result] Guo W, Li M, Dong Y, Zhou H, Zhang Z, Tian C, Qin R, Wang H, Shen Y, Du K, Zhao L, Fan H, Luo S, Hu D. Diabetes is a risk factor for the progression and prognosis of COVID-19. Diabetes Metab Res Rev. 2020 Oct;36(7):e3319. doi: 10.1002/dmrr.3319. Epub 2020 Apr 7. PMID 32233013
- [Result] Kassir R. Risk of COVID-19 for patients with obesity. Obes Rev. 2020 Jun;21(6):e13034. doi: 10.1111/obr.13034. Epub 2020 Apr 13. No abstract available. PMID 32281287
- [Result] Huespe I, Carboni Bisso I, Di Stefano S, Terrasa S, Gemelli NA, Las Heras M. COVID-19 Severity Index: A predictive score for hospitalized patients. Med Intensiva (Engl Ed). 2020 Dec 29;46(2):98-101. doi: 10.1016/j.medin.2020.12.001. Online ahead of print. No abstract available. PMID 33478781
- [Result] Prokop M, van Everdingen W, van Rees Vellinga T, Quarles van Ufford H, Stoger L, Beenen L, Geurts B, Gietema H, Krdzalic J, Schaefer-Prokop C, van Ginneken B, Brink M; COVID-19 Standardized Reporting Working Group of the Dutch Radiological Society. CO-RADS: A Categorical CT Assessment Scheme for Patients Suspected of Having COVID-19-Definition and Evaluation. Radiology. 2020 Aug;296(2):E97-E104. doi: 10.1148/radiol.2020201473. Epub 2020 Apr 27. PMID 32339082
- [Result] Moftakhar L, Moftakhar P, Piraee E, Ghaem H, Valipour A, Azarbakhsh H. Epidemiological characteristics and outcomes of COVID-19 in diabetic versus non-diabetic patients. Int J Diabetes Dev Ctries. 2021 Jul;41(3):383-388. doi: 10.1007/s13410-021-00930-y. Epub 2021 Feb 9. PMID 33584062